CLINICAL TRIAL: NCT05971420
Title: Virtual Reality Activity-based Training for Preventing Falls Among Community-dwelling Older Adults With Mild Cognitive Impairment: A Pilot Randomized Control Trial Study
Brief Title: Virtual Reality Activity-based Training for Preventing Falls for Older Adults With Mild Cognitive Impairment
Acronym: MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Queensland (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: USQ AEC H21REA071
Record Dates: First submitted 2023-07-08; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Mild Cognitive Impairment; Fall Prevention; Virtual Reality; Exercise Training
Keywords: Fall risk; VR; MCI; Ageing
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): VR activity-based training
  Interventions: Other: VR activity-based
- Exercise group (Active Comparator): Exercise-based training (Baduanjin)
  Interventions: Other: Exercise-based (Baduanjin)

INTERVENTIONS:
Other: VR activity-based — VR games activities were chosen for simulated cognitive-motor training in the VR group. The VR training modules for this study included fire drill, walking exercise, balancing game activities and community shopping practices. These training modules involved dual task components; the participant was expected to train up his/her physical and cognitive motor performances in an 8-week VR activity-based program. VR group participants received 2-sessions per week, 16 training sessions in total.
  Arms: VR group
Other: Exercise-based (Baduanjin) — The exercise group used a traditional Chinese Qigong Baduanjin exercise incorporating with a fall prevention education strategy.
  Arms: Exercise group

SUMMARY:
Using a Virtual Reality (VR) games-based application is as an innovative falls prevention technology in an aged care service. The VR intervention has promising effects on improving the physical and balance performances in the older adults.The study explored and evaluated the effects of VR activity-based training on falls prevention among community-dwelling older adults with mild cognitive impairment.

DETAILED DESCRIPTION:
A pilot randomized control trial study was applied to compare the effects on falls prevention between participants who experienced a full-immersive VR training and group-based exercise (Baduanjin) training. Eighteen participants were recruited from ausing convenience sampling and were randomly assigned into the VR group and the exercise group (non-VR). The participants in both wo groups' participants attended 16 falls prevention training sessions over eight weeks. Eligible participants identified with a higher risk of mild cognitive impairment and early dementia undertook three measurements, pretest (T1), post-test (T2) and follow up (T3). The primary outcomes assessed included changes in physical risks factor of falls, and the secondary outcomes assessed included changes in cognition and fall efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. aged 65 years to 85 years inclusive;
2. had a history of a fall within the past 2 years;
3. community-dwelling older adults;
4. at a higher risk of mild cognitive impairment and dementia, assessed by a validated screening tool of Hong Kong Montreal Cognitive assessment test (HK-MoCA score=21/22);
5. walk independently e.g. able to access publicly - VR research center centre or local community aged care facilities.

Exclusion Criteria:

if they had a medical diagnosis of unstable health conditions

1. dizziness;
2. Meniere's disease;
3. Epilepsy;
4. Parkinson's disease;
5. Severe hearing impairment and visual impairments;
6. Mental illness.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Berg balance test (BBS) - change is being assessed | At prettest, postest (up to 8 weeks) and post 3 months follow up
  To test the balance performance and assess the fall risk. Total score is 56 ( score below 51 indicated predictive of fall risk)
Time up and go test (TUG) - change is being assessed | At prettest, postest (up to 8 weeks) and post 3 months follow up
  To assess functional mobility and assess the fall risk. Score over 12 seconds indicates higher risk of fall for the older adults
Six minutes walk test (6MWT) - change is being assessed | At prettest, postest (up to 8 weeks) and post 3 months follow up
  To assess the walking speed and performance. Walking distance within 6 minutes measured the length (m/metre)

SECONDARY OUTCOMES:
Cognitive status assessed by Montreal Cognitive Assessment Scale- change is being assessed | At prettest, postest (up to 8 weeks) and post 3 months follow up
  To assess the cognitive level. Total score 30 ( score if less than 22 indicated higher risk of midl cognitive impairment
Executive functioning tests by Trail making test A and test B *TMTA/B) - change is being assessed | At prettest, postest (up to 8 weeks) and post 3 months follow up
  To assess the level of executive functions. It indicated the time of completion (second)
Fall efficacy by fall efficacy international scale (FESI) - change is being assessed | At prettest, postest (up to 8 weeks) and post 3 months follow up
  To assess the level of fear concern. Totoal score is 64 (score lower than 27 indicated less fear concern

CONTACTS AND LOCATIONS:
Overall Officials: WING KEUNG IP, Principal Investigator — University of Southern Queensland
Locations (1):
- The Hong Kong Polytechnic University, St. James Settlement Hong Kong, Salvation Army Hong Kong, Hong Kong, China, Hong Kong

IPD SHARING:
Plan to Share IPD: No
No permission from participants